CLINICAL TRIAL: NCT02109315
Title: Vitamin C and Liraglutide Effects on Hypoglycemia-induced Oxidative Stress, Inflammation and Endothelial Dysfunction in Type 1 Diabetes.
Acronym: DIAB-01
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAB-01
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2014-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide endovenous 6 mg (Experimental): Liraglutide endovenous de 0.6 mg. one time a day
  Interventions: Drug: Liraglutide 6 mg
- Vitamine C (Experimental): C Vitamine endovenous 1000 mg/5 ml. Infusion dose: 30 mgr/min
  Interventions: Drug: Vitamine C

INTERVENTIONS:
Drug: Vitamine C — C Vitamine endovenous 1000 mg/5 ml. Infusion dose: 30 mgr/min
  Arms: Vitamine C
Drug: Liraglutide 6 mg — Liraglutide endovenous de 0.6 mg. one time a day
  Arms: Liraglutide endovenous 6 mg

SUMMARY:
To investigate the effect of liraglutide on vascular injury induced hypoglycemia in patients with type 1 diabetes mellitus. The vascular damage is evaluated at investigating the changes of endothelial function

DETAILED DESCRIPTION:
To investigate the effect of antioxidants (Vitamin C) on the vascular damage induced hypoglycemia in patients with type 1 diabetes. The vascular injury was evaluated in the same way as main objective. Checking the existence of a peripheral response to the action of GLP-1 due to oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Informed and signed consent obtained before any trial-related activity . ( Trial-related activities are those procedures that were not performed during routine medical examination of the patient) .
* Diagnosis of type 1 diabetes.
* Patients who do not have autonomic dysfunction , defined by ( 1).
* Patients not showing episodes of hypoglycemia unawareness based on the methods of Gold et al (2) .
* Patients without microvascular complications of diabetes.
* Patients without macrovascular complications of diabetes.
* Patients treated with multiple daily injections of insulin.
* No smoking .
* They should have a complete blood count, lipid profile, liver profile , renal profile and plasma electrolyte levels within normal values .
* No subject must have a history of hypertension or taking medication for high blood pressure .
* No subject should be taking medications known to affect the neuroendocrine responses to hypoglycemia or anti inflammatory

Exclusion Criteria:

* Known or suspected hypersensitivity to study some related products.
* Fertile women, lactating or pregnant, intend to become pregnant or who are not using adequate contraception, or men who have sexually active and are not sterilized surgically, those whose partners are not using a method adequate contraception.
* Clinical diagnosis of Type 2 Diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Endothelial dysfunction (Flow mediated dilation): Endothelial function is assessed measuring flow-mediated vasodilation (FMD) of the brachial artery. | 8 weeks

SECONDARY OUTCOMES:
Oxidative stress markers | 8 weeks
  Oxidative stress markers (nitrotyrosine and 8-iso prostaglandin F2 alpha plasma) in serum1 inflammation markers (serum sICAM-1, interleukin 6) 1

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ceriello A Ceriello, MD, Principal Investigator — Hospital clínic i provincial de Barcelona
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain